CLINICAL TRIAL: NCT07342556
Title: EMIT-2b: Evaluating Modes of Influenza Transmission Through the Conduct of Controlled Human Influenza Virus Infection Transmission Trials (CHIVITTs)
Brief Title: Evaluating Modes of Influenza Transmission 2b Baseline SAR
Acronym: EMIT-2b-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Donald K. Milton, Distinguished University Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2313702-Baseline-SAR; U19AI162130 (NIH)
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Influenza (Healthy Volunteers)
Keywords: influenza; airborne transmission; infection transmission; touch transmission; spray (droplet) transmission
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Healthy people "Recipients" will be exposed to people who have recently become naturally infected with influenza virus in a controlled environment designed to maximize all major routes of respiratory viral infection transmission (touch contact, spray direct deposition (previously called droplet), and airborne-inhalation transmission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure to Donors with naturally acquired influenza infection under controlled conditions (Other): Recipients are exposed to Donors in a controlled environment while performing prescribed activities, including playing cards and other games, and periodically shaking hands with Donors and rubbing their own nose and eyes.
  Interventions: Other: Exposure to Donors with naturally acquired influenza virus infection

INTERVENTIONS:
Other: Exposure to Donors with naturally acquired influenza virus infection — Recipients are exposed to Donors in a controlled environment while performing prescribed activities, including playing cards and other games, and periodically shaking hands with Donors and rubbing their own nose and eyes.

SUMMARY:
This is a research study to investigate how influenza transmits from person-to-person. Participation as a healthy "Recipient" in this study involves:

* Home semi-quarantine lasting about 14 days during which the participants must wear an N95 in class and take other precautions
* Daily assessments and clinic visits for 14 days
* Spending every weekday evening for about 14 days from around 6 - 10 pm, including a provided dinner, in a controlled environment. There may be additional sessions and different required participation times on weekends
* Exposure to people infected with influenza in the controlled environment
* Three blood draws, at the start, at the end of 14 days, and about a month after the end.
* A follow-up clinic visits one month after the end of home semi-quarantine
* A two-month follow-up phone call. This study may increase the participant's risk of catching influenza.

If the participants get infected during the study, the investigators may:

* Provide the participants with a prescription for antiviral medication or
* Refer the participants for medical care
* Ask the participants to become a Donor and expose other Recipients.

The participants will be compensated for their time and active participation in the study; however, they may not personally benefit from the study. While the participants may receive supportive care for an infection resulting from the study, this is not meant to replace their regular medical care. If the participants become very ill and need referral for medical care, they or their medical insurance will be billed.

If the participants are someone who recently became infected with influenza either through their daily activities or by participating in this study as a Recipient, they are invited to participate in this research study as a Donor and interact with a group of health participants in a controlled environment. Participation in this study as a Donor involves exposing Recipients for at least one and up to five days including:

* Attend exposure events in a controlled environment

  * Weekday evenings from around 6-10 pm
  * Additional day and evening events on weekends
  * Events include a provided dinner
* Daily assessments and clinic visits for 1 to 5 days
* Provide exhaled breath samples for 30 to 60 minutes
* Three blood draws, at the start and end of exposure events, and about a month after the end
* A follow-up clinic visit one month after their last exposure event
* A two-month follow-up phone call

If the participants experience severe symptoms related to their influenza infection, we may:

* Provide the participants with a prescription for antiviral medication or
* Refer the participants for medical care

The participants will be compensated for their time and active participation in the study; however, they may not personally benefit from the study. While the participants may receive supportive care for their influenza infection, this is not meant to replace their regular medical care. If the participants become very ill and need referral for medical care, they or their medical insurance will be billed.

ELIGIBILITY:
Inclusion Criteria Recipients:

1. Enrolled in the Recipient Registry (UMD IRB Protocol # 2303473, eligible age ≥18 and ≤49)
2. Provides written informed consent, can comply with the planned study procedures, is available for an up to ~14-day home semi-quarantine period, and can attend scheduled exposure events and scheduled follow-up visits.
3. Participants must be able to comprehend the study requirements, as evidenced by a score of 100% on the comprehension assessment (repeated tries permitted).
4. No significant change (for the worse) in general health history or in concomitant medication use, as compared from their responses collected during screening (Recipient Protocol).
5. Live in a private, single occupancy bedroom and agree to take precautions to avoid contracting a respiratory infection outside of the controlled exposure events through a home semi-quarantine prescribed by investigators.
6. Agree not to meet with other participants (Recipients or Donors) outside of the programmed exposure events during their participation in the home semi-quarantine.

Exclusion Criteria Recipients:

1. Female of childbearing potential who has a positive urine pregnancy test within 24 hours of enrollment in a Recipient Cohort or is breastfeeding or planning to become pregnant within 2 months after enrollment.
2. Presence of infection with influenza, SARS-CoV-2, or other respiratory pathogens detected via a multiplex nucleic acid amplification test (e.g., TaqMan Array Card assay) at entry to the transmission trial.

   a. Volunteers with influenza infection may be eligible to enroll as Donors.
3. Within the past 72 hours, presence of influenza-like illness, as defined as fever of ≥100.2°F AND cough or sore throat, in the absence of an alternative cause.
4. Receipt of any blood products within the past 2 months.
5. Does not agree to provide permission for secondary research use of extra samples collected and stored specimens.
6. Habitual smoker of tobacco, marijuana, or e-cigarettes per self-report. (Habitual smokers are those who smoke or vape more than four cigarettes, other tobacco products, e-cigarettes or marijuana in a week for more than three months or use an inhaled nicotine or marijuana product more than 3 days a week on average. Edible or patch forms of tobacco or marijuana products do not constitute an exclusion.)
7. Self-reported or known history of alcohol or drug abuse in the past two years and/or illicit drug use within the last 30 days. (Prescribed stimulants for the treatment of ADHD and cannabinoids use do not constitute exclusionary criteria)
8. Has an ongoing symptomatic condition for which the individual has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan. (symptomatic condition means for example ongoing chronic fatigue without a diagnosis for symptom.)
9. Presence of self-reported or medically documented significant medical or psychiatric condition(s) Significant medical or psychiatric conditions include but are not limited to:

   1. Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma, cystic fibrosis) requiring daily medications* currently or any treatment of respiratory disease exacerbations or hospitalizations for acute respiratory illnesses (e.g., asthma exacerbation) in the last 5 years. (* Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.)
   2. Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
   3. Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).
   4. Ongoing malignancy or recent diagnosis of malignancy, including leukemia; treated, non-melanoma skin cancers are permissible.
   5. An autoimmune disease.
   6. An immunodeficiency of any cause.
   7. A blood disorder (e.g., sickle cell disease)
   8. Endocrine disorders (e.g., diabetes)
   9. Liver, kidney, metabolic disorders
   10. BMI ≥40 kg/m2
   11. Persistent post-viral syndromes with ongoing cardiovascular, respiratory, or neurologic conditions.
   12. Any other condition or behavior that in the opinion of the PI would affect the ability to participate in the screening or future transmission studies.
10. Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness. Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 2-month period. Low dose topical and intranasal steroid preparations used for a discrete period are permitted.
11. Known allergy or intolerance to treatments for influenza and other respiratory infections (including but not limited to oseltamivir, baloxavir, acetaminophen/paracetamol).
12. History of a previous severe allergic reaction to medicines of any kind with generalized urticaria, angioedema, or anaphylaxis.
13. Participating in any other interventional clinical trial that has a scheduled intervention 30 days prior to the start or after the end of the home semi-quarantine.

Inclusion Criteria Donors:

1. Provides written informed consent, able to comply with the planned study procedures, available for between 1 and 5 days of multiple hour daily transmission experiments in a controlled environment research facility for the transmission trial and can attend the scheduled follow-up visits.
2. Comprehends the study requirements, as evidenced by a score of 100% on the comprehension assessment (repeated tries permitted).
3. Males and non-pregnant, non-breastfeeding females1 aged ≥18 and ≤59 years of age, at time of initial consent. Pregnancy and breastfeeding status to be determined by self-report.
4. Agrees to the collection of specimens for secondary research.
5. Evidence of onset of respiratory infection within the past 48 hours at time of entry into the Donor's initial exposure event, including one or more of the following:

   1. Onset of influenza-like illness, as defined as fever (measured oral temperature of ≥100.2°F or self-reported fever in the absence of a measured temperature) AND cough or sore throat in the setting of local influenza activity.
   2. Onset of less specific symptoms with a positive molecular test for influenza virus infection.
   3. Laboratory-confirmed influenza infection (including rapid antigen test in the setting of known local influenza activity) with significant exposure to a laboratory confirmed influenza case (e.g., a roommate) within the last 4 days in the absence of symptoms.

Exclusion Criteria Donors:

1. Female of childbearing potential who is breastfeeding or has positive urine pregnancy test upon enrollment.
2. Presence of self-reported or medically documented significant medical or psychiatric condition(s) Significant medical or psychiatric conditions include but are not limited to:

   1. Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma, cystic fibrosis) requiring daily medications currently or any treatment of respiratory disease exacerbations or hospitalizations for acute respiratory illnesses (e.g., asthma exacerbation) in the last 5 years. Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.
   2. Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
   3. Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).
   4. Ongoing malignancy or recent diagnosis of malignancy, including leukemia; treated, non-melanoma skin cancers are permissible.
   5. An autoimmune disease.
   6. An immunodeficiency of any cause.
   7. A blood disorder (e.g., sickle cell disease)
   8. Endocrine disorders (e.g., diabetes)
   9. Liver, kidney, metabolic disorders
   10. BMI ≥40 kg/m2
   11. Persistent post-viral syndromes with ongoing cardiovascular, respiratory, or neurologic conditions.
   12. Any other condition or behavior that in the opinion of the PI would affect the ability to participate in the transmission study over the next several days.
   13. Meets criteria for escalation of care at the time of enrollment visit (will be referred for care).
3. Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 2-month period. Low dose topical and intranasal steroid preparations used for a discrete period are permitted.
4. Ongoing symptomatic condition for which individual has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan.

   e.g., ongoing and debilitating fatigue without a diagnosis for the symptom.
5. Self-reported or known history of alcohol or drug abuse within the past two years or illicit drug use within the last 30 days.
6. Is a habitual smoker of tobacco, marijuana, or e-cigarettes per self-report. Habitual smokers are those who smoke or vape more than four cigarettes, other tobacco products, e-cigarettes or marijuana in a week for more than three months or use an inhaled nicotine or marijuana product more than 3 days a week on average. Edible or patch forms of tobacco or marijuana products do not constitute an exclusion.
7. Known allergy or intolerance to treatments for influenza and other respiratory infections (including but not limited to acetaminophen/paracetamol).
8. History of a previous severe allergic reaction to medicines of any kind with generalized urticaria, angioedema, or anaphylaxis.
9. Presence of infection with SARS-CoV-2, as detected via a multiplex nucleic acid amplification test (e.g., Cepheid 4-Plex).
10. Participating in any other interventional clinical research study that has a scheduled intervention 30 days prior to or after the transmission trial.
11. Any condition, to include medical and psychiatric conditions, that in the opinion of the Investigator, might interfere with the safety of the participant or the study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PCR confirmed transmission of influenza virus infection | 1 month
  Transmission of influenza infection defined as having >1 nasal swab test positive for an influenza virus matching the type and subtype detected in a trial Donor.
Genomic sequencing-confirmed transmission of influenza virus infection | 1 month
  Sequencing-confirmed transmission will be defined as a Recipient infection with a virus having ≤2 nucleotide difference from the virus infecting a trial Donor and closer genetic relationship to the apparent source Donor than Donors recruited from the community are to each other.
Culture-confirmed transmission of influenza virus infection | 1 month
  Culture-confirmed transmission will be defined as positive viral culture for a virus that is also a sequence match to a virus cultured from a Donor.

CONTACTS AND LOCATIONS:
Overall Officials: Donald K Milton, MD, DrPH, Principal Investigator — University of Maryland School of Public Health
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available through appropirate repositories (e.g. OSF.io) using REDCap's de-identification options. REDCap is a HIPAA compliant data system which we will use to store data and distribute electronic informed consent forms and surveys. This system provides de-identification options that we can use to generate de-identified data by removing known identifier fields, invalidated text fields, notes fields, and/or date fields. We can also use it to shift date and/or hash record names so the actual values will be hidden.
Time Frame: IPD will be made publicly available at the time of publication of study results and will be published in a permanent (to the extent that the internet is permanent) repository with permanent DOI.
Access Criteria: Publicly available via a DOI included in publications.

REFERENCES:
- [Background] Nguyen-Van-Tam JS, Killingley B, Enstone J, Hewitt M, Pantelic J, Grantham ML, Bueno de Mesquita PJ, Lambkin-Williams R, Gilbert A, Mann A, Forni J, Noakes CJ, Levine MZ, Berman L, Lindstrom S, Cauchemez S, Bischoff W, Tellier R, Milton DK; EMIT Consortium. Minimal transmission in an influenza A (H3N2) human challenge-transmission model within a controlled exposure environment. PLoS Pathog. 2020 Jul 13;16(7):e1008704. doi: 10.1371/journal.ppat.1008704. eCollection 2020 Jul. PMID 32658939
- [Background] Lai J, Sobhani H, Coleman KK, Tai SS, Hong F, Sierra Maldonado I, Esparza Y, McPhaul KM, Zhu S, DeVoe DL, Ortiz JR, Chen S, Yellin T, Carreno JM, Krammer F, Cowling BJ, Gordon A, Chen WH, Srebric J, Milton DK; EMIT-2 Study Team. Evaluating modes of influenza transmission (EMIT-2): Insights from lack of transmission in a controlled transmission trial with naturally infected donors. PLoS Pathog. 2026 Jan 7;22(1):e1013153. doi: 10.1371/journal.ppat.1013153. eCollection 2026 Jan. PMID 41499634
- See also: A link for information about volunteering as a healthy participant — https://sites.google.com/umd.edu/phablabumd/emit-2b